CLINICAL TRIAL: NCT03316209
Title: Identification of Occupational Exposures in Acute Hematologic Malignancy
Acronym: RHELYPRO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: ANSES (Other)
Responsible Party: Sponsor
Other Study IDs: RHELYPRO
Record Dates: First submitted 2017-08-01; First posted 2017-10-20 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Non Hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Multiple Myeloma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lymphoid hemopathies are a group of malignant haematological disorders characterized by clonal proliferation of cells of the lymphoid line. Non-Hodgkin's lymphoma (NHL), chronic lymphocytic leukemia (CLL), and multiple myeloma (MM) are the most frequently encountered features of lymphoid hemopathies. Duriong the last 35 years the prevalence of these pathologies has increased in France but also in most industrialized countries. This increased can't be solely explained by demographic changes and improvements in diagnostic techniques. As a result, the involvement of environmental and professional factors is strongly suspected. Studies have shown that these diseases are associated with some professions or type of activity, including agricultural occupations, and other sectors such as agriculture, printing, woodworking. Some organic solvents and pesticides have been suspected of being risk factors of hematologic malignancies. Based on cohort studies and case-control studies, some of them have been identified by the International Cancer Research Center as associated with the occurrence of NHL with a sufficient or limited level of evidence. One of the difficulties encountered in the analysis of the literature has been the permanent evolution of the international classification of lymphoid hemopathies over the past 30 years. The old epidemiological studies are therefore difficult to interpret. Lymphoid hemopathies cover a range of different conditions, thus it is likely that carcinogens involved vary according to the type of hemopathy. Finally, environmental and occupational exposures to various chemicals and biological agents have evolved over time. The aim of this study is firstly to develop and validate a questionnaire to identify and quantify exposures to nuisances (substances and agents) suspected of being associated with the occurrence of NHL, MM and LLC. In a second time, this questionnaire will be used as a support for the realization of a subsequent case-control study to improve epidemiological knowledge on these diseases.

DETAILED DESCRIPTION:
This study is a prospective, multicenter study on patients with a diagnosis of NHL, MM or CLL. All the patients with a diagnosis of NHL, MM or CLL in the participant centers will be purposed to participate. Each patient included will have an interview with a clinical study technician or doctor of occupational medicine. A specific detailed questionnaire has been created for the study. It focuses on specialized professional careers to spread occupational exposures to nuisances (substances and agents) suspected of being associated with NHL, MM or LLC risk. Each questionnaire will be evaluated by a physician expert in occupational disease, to conclude on the parameters exposure to the various suspected carcinogens. The study will cover 300 patients.

ELIGIBILITY:
Inclusion Criteria:

* Incident cases of NHL, MM and CLL diagnosed in hospital hematology departments participating in the study.
* Age between 20 and 80 years

Exclusion Criteria:

* HIV infection
* History of organ or marrow transplant

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be proposed to all the patients diagnosed with NHL, MM and CLL aged between 20 and 80 years old, without HIV infection and history of bone marrow transplant. If the patients agree to participate, a clinical research technician or a physician will give them a 2-hour questionnaire on their past occupational and exposures to toxic products. This filled questionnaire will then be interpreted by a specialized doctor to evaluate the exposition to each toxic products.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
ability of the questionnaire to identify occupational carcinogenic exposures | day 1
  included patient will complete a questionnaire (duration: 2 hours). this questionnaire will be interpreted by an expert physician in occupational diseases

SECONDARY OUTCOMES:
Acceptability of the questionnaire by patients | day 1
Determination of the number of subjects recorded as suffering of an occupational disease | day 1
Professional sectors concerned by each nuisance | day 1
Activities concerned by each nuisance | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Murielle GAIN, MD, Principal Investigator — Centre Hospitalier intercommunal de Créteil
Locations (7):
- France (7):
  - CHU Bordeaux, Bordeaux
  - CHU Caen, Caen
  - CHU H. Mondor, Créteil
  - Service de pathologie professionelle, Créteil
  - CHRU Lille, Lille
  - Fernand Widal hospital, Paris
  - CHU Toulouse, Toulouse